CLINICAL TRIAL: NCT05190211
Title: The Effectiveness of Synchronized Online and Video-based Exercise Programs in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Telerehabilitation in Patients With Idiopathic Pulmonary Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPFTele
Record Dates: First submitted 2021-11-26; First posted 2022-01-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-04

CONDITIONS: IPF
Keywords: IPF; telerehabilitation; videobased rehabilitation; exercise; physical therapy; pulmonary rehabilitation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The cases meeting the inclusion criteria will be randomized and divided into two groups, the groups will be named as Telerehabilitation Exercise Group (TGr) and Video Group (VGr).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (TG) (Experimental)
  Interventions: Other: Telerehabilitation exercise program
- Video Group (VGr) (Experimental)
  Interventions: Other: Videobased exercise program

INTERVENTIONS:
Other: Telerehabilitation exercise program — TGr will be given online exercises, synchronized 2 days a week, and a home program for 1 day, accompanied by a physiotherapist, via videoconference on the group smartphone.
  Arms: Telerehabilitation Group (TG)
Other: Videobased exercise program — After 1 session of online simultaneous exercise training in the company of a physiotherapist via videoconference on the smart phone, an exercise video including the exercises will be sent to them and the patients will be asked to do their exercises 3 days a week. The subjects will be asked to keep an exercise diary and the status of the diaries will be followed by calling them once a week.
  Arms: Video Group (VGr)

SUMMARY:
It is to determine the effectiveness of different telerehabilitation exercise programs received to 2 groups randomly formed in idiopathic pulmonary fibrosis (IPF) patients. The cases meeting the inclusion criteria will be randomized and divided into two groups, the groups will be named as Telerehabilitation Exercise Group (TGr) and Video Group (VGr).

DETAILED DESCRIPTION:
Patients diagnosed with idiopathic pulmonary fibrosis by a chest diseases specialist and referred to pulmonary rehabilitation will be included in the study. The cases meeting the inclusion criteria will be randomized and divided into two groups, the groups will be named as Telerehabilitation Exercise Group (TGr) and Video Group (VGr). TGr will be given online exercises, synchronized 2 days a week, and a home program for 1 day, accompanied by a physiotherapist, via videoconference on the group smartphone. As for the VGr group, after 1 session of online simultaneous exercise training in the company of a physiotherapist via videoconference on the smart phone, an exercise video including the exercises will be sent to them and the patients will be asked to do their exercises 3 days a week. The subjects will be asked to keep an exercise diary and the status of the diaries will be followed by calling them once a week. The exercise period will be 8 weeks for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-75
* Having a diagnosis of IPF disease diagnosed according to the following clinical diagnostic criteria according to the American Thoracic and European Respiratory Societies (ATS-ERS)
* Presence of dyspnea on exertion
* Stable clinical state at the time of admission without infection or exacerbation in the previous 4 weeks

Exclusion Criteria:

* Patients with severe comorbid diseases, unstable coronary artery disease, collagen vascular diseases and needing high flow oxygen therapy (˃ 3-4 L \min).
* A history of effort-related syncope or any comorbidity (such as severe orthopedic or neurological deficits or unstable heart disease) that precludes exercise training.
* Participation in a pulmonary rehabilitation program within the past 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The exercise capacity | Change from baseline 6 minute walking distance at 8 weeks
  The exercise capacity will be assessed by the 6 minute walking test.The test was conducted in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines.

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | Change from baseline FVC at 8 weeks
  Forced vital capacity will be assessed by the spirometer. Pulmonary function test will performe by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines
Perception of dyspnea | Change from baseline dyspnea perception at 8 weeks
  Perception of dyspnea will be evaluated by Modified Medical Research Council Dyspnea scale. The mMRC Dyspnea Scale is best used to establish baseline functional impairment due to dyspnea attributable to respiratory disease; tracking the mMRC over time or with therapeutic interventions is of less certain clinical utility.The severity of dyspnea is rated on a scale of 0 to 4. "O" means no dyspnea perception, "4" means severe dyspnea perception.
Respiratory muscle strength | Change from baseline respiratory muscle strength at 8 weeks
  Respiratory muscle strength will be evaluated by the intraoral pressure measurement device.The mouth pressure measurement was performed with the Cosmed Pony Fx. Patient placed a rubber mouthpiece with flanges, on the device, sealed their lips firmly around the mouthpiece, exhaled/inhaled slowly and completely, and then tried to breath in as hard as possible. The patient was allowed to rest for about a minute and the maneuver was repeated five times. Verbal or visual feedback was provided after each maneuver. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value was obtained.
Peripheral muscle strength | Change from baseline peripheral muscle strength at 8 weeks
  Peripheral muscle strength will be assessed by the hand held dynamometer
Perception of general fatigue | Change from baseline perception of general fatigue at 8 weeks
  Perception of fatigue will be assessed by the Fatigue severity scale.The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity. Another way of scoring: mean of all the scores with minimum score being 1 and maximum score being 7.
Saint George Respiratory Questionnaire (SGRQ) score | Change from baseline SGRQ score at 8 weeks
  The quality of life will be assessed by the Saint George Respiratory Questionnaire.The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life)
Hospital anxiety and depression scale score | Change from baseline anxiety level at 8 weeks
  The anxiety levels will be evaluated by Hospital anxiety and depression scale.The total score ranges from 0-63. The following guidelines are recommended for the interpretation of scores: 0-9, normal or no anxiety; 10-18, mild to moderate anxiety; 19-29, moderate to severe anxiety; and 30-63, severe anxiety.
International Physical Activity Questionnaire- short form | Change from baseline physical activity level at 8 weeks
  Physical activity level will be assessed by International Physical Activity Questionnaire- Short form. Including seven questions on the frequency and duration of time spent in physical activity in the past 7 days to calculate a score for each domain (walking, moderate-intensity activities and vigorous-intensity activities) and an overall grand total expressed in MET-minutes/week.MET values and Formula for computation of Met-minutes Walking MET-minutes/week = 3.3 * walking minutes * walking ëdaysí Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days A combined total physical activity MET-min/week can be computed as the sum of Walking + Moderate + Vigorous MET-min/week scores.
Forced expiratory volume in one second (FEV1) | Change from baseline FEV1 at 8 weeks
  Forced expiratory volume in one second will be assessed by the spirometer. Pulmonary function test will performe by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided